CLINICAL TRIAL: NCT05186285
Title: A Single-dose, Randomized, Double Blind, Placebo-controlled, Dose-increasing Study to Evaluate the Safety, Tolerability, PK Characteristics, PD Effect, and Immunogenicity of CM338 Injection in Healthy Subjects.
Brief Title: Single Ascending Dose Study of CM338 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM338HV001
Record Dates: First submitted 2021-11-23; First posted 2022-01-11 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- CM338 30mg, IV (Experimental): 30mg, single dose, IV
  Interventions: Drug: CM338
- CM338 60mg, IV (Experimental): 60mg, single dose, IV
  Interventions: Drug: CM338
- CM338 120mg, IV (Experimental): 120mg, single dose, IV
  Interventions: Drug: CM338
- CM338 240mg, IV (Experimental): 240mg, single dose, IV
  Interventions: Drug: CM338
- CM338 240mg, SC (Experimental): 240mg, single dose, SC
  Interventions: Drug: CM338
- CM338 480mg, IV (Experimental): 480mg, single dose, IV
  Interventions: Drug: CM338
- CM338 600mg, IV (Experimental): 600mg, single dose, IV
  Interventions: Drug: CM338
- CM338 600mg, SC (Experimental): 600mg, single dose, SC
  Interventions: Drug: CM338
- Placebo (Placebo Comparator): Placebo, single dose, IV or SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM338 — CM338 : a humanized monoclonal antibody.
  Arms: CM338 120mg, IV; CM338 240mg, IV; CM338 240mg, SC; CM338 30mg, IV; CM338 480mg, IV; CM338 600mg, IV; CM338 600mg, SC; CM338 60mg, IV
Drug: Placebo — Placebo.
  Arms: Placebo

SUMMARY:
This study was a single-center, randomized, double blind, placebo-controlled, single-dose, dose-increasing study to evaluate the safety, tolerability, PK characteristics, PD effect, and immunogenicity of CM338 injection administered intravenously or subcutaneously at different doses in healthy subjects.

DETAILED DESCRIPTION:
The study included screening period, baseline period, administration and hospitalization observation period, and safety follow-up period.

Sixty-six healthy volunteers will be enrolled and randomized into 8 groups.

ELIGIBILITY:
Inclusion Criteria:

* with the ability to understand this study and voluntarily sign the informed consent form.
* 18 to 65 years of age.
* with normal or abnormal without clinically significance on medical history, vital signs, physical examination, 12-lead ECG, laboratory examination, chest X-ray, and abdominal color ultrasound, etc.
* able to communicate with the researchers and follow the requirements specified in the protocol.
* agree to use effective contraceptive methods from signing the ICF to 6 months after the administration.

Exclusion Criteria:

* plan to conduct any major surgery during the study.
* known allergy to monoclonal antibody drugs or other related drugs, or to the excipients of CM338 injection.
* with any clinical history including serious diseases or circulatory system, endocrine system, nervous system, blood system, immune system, mental system and metabolic abnormalities.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Safety : Incidence of Adverse Events (AEs). | Baseline up to Day 57
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter : Peak Plasma concentration (Cmax) | Baseline up to Day 57
  Peak Plasma concentration (Cmax)
Pharmacokinetics (PK) parameter : Time to reach peak concentration (Tmax) | Baseline up to Day 57
  Time to reach peak concentration (Tmax)
Pharmacokinetics (PK) parameter : Area under the plasma concentration-time curve from 0 to ∞ (AUC0-∞) | Baseline up to Day 57
  Area under the plasma concentration-time curve from 0 to ∞ (AUC0-∞)
Pharmacokinetics (PK) parameter : Area under the plasma concentration-time curve from 0 to t (AUC0-t) | Baseline up to Day 57
  Area under the plasma concentration-time curve from 0 to t (AUC0-t)
Pharmacokinetics (PK) parameter : Clearance rate (CL/F) | Baseline up to Day 57
  Clearance rate (CL/F)
Bioavailability : bioavailability of CM338 with SC | Baseline up to Day 57
  The bioavailability of CM338 with SC
Pharmacodynamics (PD) : C4b deposition activity of mannose-binding lectin serine protease 2 (MASP-2) in serum. | Baseline up to Day 57
  C4b deposition activity of mannose-binding lectin serine protease 2 (MASP-2) in serum.
Pharmacodynamics (PD) : the content of mannose-binding lectin serine protease 2 (MASP-2) in serum. | Baseline up to Day 57
  The content of mannose-binding lectin serine protease 2 (MASP-2) in serum.
Immunogenicity: Proportion of subjects with anti-drug antibody (ADA). | Baseline up to Day 57
  Proportion of subjects with anti-drug antibody (ADA).

CONTACTS AND LOCATIONS:
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China